CLINICAL TRIAL: NCT02886156
Title: Effects of Continuous Positive Airway Pressure on Cognitive Function, Neurocognitive Architecture and Function in Patients With Obstructive Sleep Apnea: The Shanghai Multicenter Obstructive Sleep Apnea Therapy Trial
Brief Title: Effects of CPAP on Cognitive Function, Neurocognitive Architecture and Function in Patients With OSA: The SMOSAT Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Huajun Xu, Residents, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6thShanghaiJiaotongU2
Record Dates: First submitted 2016-08-03; First posted 2016-09-01 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Apnea, Sleep
Keywords: OSA; CPAP; cognitive function; gut microbiota; metabolomics
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP plus BSC (Experimental): Participants in the CPAP plus BSC group will receive CPAP treatment plus the aforementioned BSC intervention. CPAP treatment (LOTUS AUTO; Curative Medical Technology Inc., Beijing, China) will be initiated using standard clinical practice at each center.
  Interventions: Device: CPAP; Dietary Supplement: BSC
- BSC intervention (Active Comparator): Participants in the BSC only group will receive advice regarding lifestyle modification, sleep hygiene, naps, exercise, caffeine, and diet, and avoiding alcohol consumption, but no specific weight loss program, diet, or salt restriction will be suggested.
  Interventions: Dietary Supplement: BSC

INTERVENTIONS:
Device: CPAP — CPAP plus BSC group Participants in the CPAP plus BSC group will receive CPAP treatment plus the aforementioned BSC intervention. CPAP treatment (LOTUS AUTO; Curative Medical Technology Inc., Beijing, China) will be initiated using standard clinical practice at each center. Participants in both groups will be asked to continue their usual medical care during the trial.
  Arms: CPAP plus BSC
Dietary Supplement: BSC — BSC only group Participants in the BSC only group will receive advice regarding lifestyle modification, sleep hygiene, naps, exercise, caffeine, and diet, and avoiding alcohol consumption, but no specific weight loss program, diet, or salt restriction will be suggested.

SUMMARY:
Multiple clinical studies have indicated that obstructive sleep apnea (OSA), the most common chronic sleep disorder, may affect neurocognitive function, and that treatment for continuous positive airway pressure (CPAP) has some neurocognitive protective effects against the adverse effects of OSA. However, the effects of CPAP treatment on neurocognitive architecture and function remain unclear. Therefore, this multicenter trial was designed to investigate whether and when neurocognitive architecture and function in patients with OSA can be improved by CPAP treatment, and to explore the role of gut microbiota in improving neurocognitive function during treatment.This study will be a multicenter, randomized, controlled trial with allocation concealment and assessor blinding. A total of 148 eligible patients with severe OSA will be enrolled from five sleep centers, and randomized to receive CPAP with best supportive care (BSC) intervention or BSC intervention alone. Cognitive function, structure and function of brain regions, gut microbiota, metabolites, biochemical variables, electrocardiography, echocardiography, pulmonary function, and arterial stiffness will be assessed at baseline before randomization and at 3, 6, and 12 months. In addition, the investigators will enroll 74 healthy controls and assess all of the aforementioned variables at baseline.

DETAILED DESCRIPTION:
Background Multiple clinical studies have indicated that obstructive sleep apnea (OSA), the most common chronic sleep disorder, may affect neurocognitive function, and that treatment for continuous positive airway pressure (CPAP) has some neurocognitive protective effects against the adverse effects of OSA. However, the effects of CPAP treatment on neurocognitive architecture and function remain unclear. Therefore, this multicenter trial was designed to investigate whether and when neurocognitive architecture and function in patients with OSA can be improved by CPAP treatment, and to explore the role of gut microbiota in improving neurocognitive function during treatment.

Methods/Design This study will be a multicenter, randomized, controlled trial with allocation concealment and assessor blinding. A total of 148 eligible patients with severe OSA will be enrolled from five sleep centers, and randomized to receive CPAP with best supportive care (BSC) intervention or BSC intervention alone. Cognitive function, structure and function of brain regions, gut microbiota, metabolites, biochemical variables, electrocardiography, echocardiography, pulmonary function, and arterial stiffness will be assessed at baseline before randomization and at 3, 6, and 12 months. In addition, the investigators will enroll 74 healthy controls and assess all of the aforementioned variables at baseline.

Ethics and Dissemination Ethics approval was given by the Medical Ethics Committee of Shanghai Jiao Tong University Affiliated Sixth People's Hospital (approval number 2015-79). The findings from this study will be disseminated in peer-reviewed journals and at conferences.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Age 30-65 years
3. Newly diagnosed OSA (full-night in-laboratory polysomnography [PSG] with AHI ≥ 15 events per hour)
4. Adherence to CPAP treatment
5. No participation in any other clinical trial in the past 3 months
6. Able to accomplish relevant tests and follow-up

Exclusion Criteria:

1. Severe systemic diseases (e.g., cardiac, hepatic, and renal failure)
2. Psychiatric conditions (e.g., depression, mania, schizophrenia)
3. Neurological diseases (e.g., head trauma, brain tumor, epilepsy, stroke, transient ischemic attack, coma)
4. Sleep disorders other than OSA (narcolepsy, insomnia, chronic sleep deprivation, rapid eye movement [REM] behavior disorder and restless legs syndrome, central sleep apnea or obesity hypoventilation syndrome)
5. Alcoholism, drug addiction, use of psychotropic drugs, sedatives, or narcotics
6. Prior therapy for OSA (i.e., CPAP, upper airway surgery, oral appliance)
7. Minimum Mental State Examination (MMSE)< 24
8. Left-handed
9. MRI contraindications (e.g., claustrophobic or metal implantation)
10. Gastrointestinal surgery during the last year, except for appendicitis and hernia surgery
11. Pregnancy
12. Use of intestinal flora regulator (e.g., antibiotics or probiotics) in the previous 8 weeks
13. Medical treatment for cholecystitis, gallstones, gastrointestinal ulcers, urinary tract infection, acute pyelonephritis, or cystitis in the past 3 months
14. Infectious diseases, such as tuberculosis, acquired immune deficiency syndrome
15. Commercial drivers or people deemed to be at risk of driving -related accidents
16. Deemed by the researchers to be suitable for this trial

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline neurocognitive function in participants at 3 month,6 month,1 year follow-up as measured by montreal cognitive assessment-score range 0-30 | baseline,month 3, month 6 and year 1
  Assessment of neurocognitive function by montreal cognitive assessment-score range 0-30

SECONDARY OUTCOMES:
Changes from baseline daytime sleepiness and sleep variables in participants at 3 month, 6 month and 1 year follow-up as measured by polysomnography (PSG) | baseline,month 3, month 6 and year 1
  Assessment of daytime sleepiness and sleep variables by PSG
Changes from baseline neurocognitive function in participants at 3 month, 6 month and 1 year follow-up as measured by central auditory processing testing | baseline,month 3, month 6 and year 1
  Assessment of neurocognitive function by central auditory processing testing
Changes from baseline neurocognitive function in participants at 3 month, 6 month and 1 year follow-up as measured by 256-channel high-density electroencephalography (EEG) recordings | baseline,month 3, month 6 and year 1
  Assessment of neurocognitive function by 256-channel high-density electroencephalography (EEG) recordings
Changes from baseline gut microbiomes in stool specimens in participants at 3 month, 6 month and 1 year follow-up as measured through metagenomic analysis | baseline,month 3, month 6 and year 1
  The bacterial genomic DNA was extracted from tool of participants,V1-V3 hypervariable regions of 16S rRNA were amplified by PCR from DNA using barcoded fusion primers,after the PCR products were extracted and quantified, they were pooled in equimolar concentrations and were sequenced using a 454 Life Sciences Genome Sequencer FLX system
Changes from baseline metabolomics profiling in participants at 3 month, 6 month and 1 year follow-up as measured by metabolomics approach | baseline,month 3, month 6 and year 1
  Metabolomics profiling will be detected by a combination of ultra-performance liquid chromatography coupled with quadrupole time-of-flight mass spectrometry (UPLC-Q-TOF-MS) and gas chromatography coupled with time-of-flight mass spectrometry (GC-TOF-MS)
Changes from baseline arterial stiffness (pulse wave velocity, ankle brachial index, toe-brachial) in participants at 3 month, 6 month and 1 year follow-up as measured by echocardiography | baseline,month 3, month 6 and year 1
  Assessment of arterial stiffness
Changes from baseline general heart function (left ventricular volume and ejection fraction)in participants at 3 month, 6 month and 1 year follow-up as measured by echocardiography | baseline,month 3, month 6 and year 1
  Assessment of general heart function
Changes from baseline body fat distribution in participants at 3 month, 6 month and 1 year follow-up | baseline,month 3, month 6 and year 1
  Assessment of body fat distribution ( abdominal subcutaneous fat,abdominal visceral fat, intrahepatic lipid) by means of magnetic resonance imaging
Changes from baseline neurocognitive function in participants at 3 month, 6 month and 1 year follow-up as measured by the neuropsychological tests. | baseline,month 3, month 6 and year 1
  The neuropsychological tests includes mental arithmetic,memory scanning, movement perception,switching attention,space location memory span,attention allocation choice reaction time curve fit
Changes from baseline Optic nerve fiber layer thickness in participants at 3 month, 6 month and 1 year follow-up as measured by optical coherence tomography | baseline,month 3, month 6 and year 1
  Assessment of Optic nerve fiber layer thickness by optical coherence tomography
Changes from baseline neurocognitive function in participants at 3 month,6 month,1 year follow-up as measured by minimum mental state examination-score range 0-30 and functional magnetic resonance imaging | baseline,month 3, month 6 and year 1
  Assessment of neurocognitive function by minimum mental state examination-score range 0-30 and functional magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Shankai Yin, MD, Ph D, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Otolaryngological Institute of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Department of Epidemiology, School of Public Health, Shanghai Jiao Tong University
Supporting Information: Study Protocol
Time Frame: After 2019
Access Criteria: Research institutions

REFERENCES:
- [Background] Henderson LA, Fatouleh RH, Lundblad LC, McKenzie DK, Macefield VG. Effects of 12 Months Continuous Positive Airway Pressure on Sympathetic Activity Related Brainstem Function and Structure in Obstructive Sleep Apnea. Front Neurosci. 2016 Mar 10;10:90. doi: 10.3389/fnins.2016.00090. eCollection 2016. PMID 27013952
- [Background] Dalmases M, Sole-Padulles C, Torres M, Embid C, Nunez MD, Martinez-Garcia MA, Farre R, Bargallo N, Bartres-Faz D, Montserrat JM. Effect of CPAP on Cognition, Brain Function, and Structure Among Elderly Patients With OSA: A Randomized Pilot Study. Chest. 2015 Nov;148(5):1214-1223. doi: 10.1378/chest.15-0171. PMID 26065720
- [Background] Rosenzweig I, Glasser M, Crum WR, Kempton MJ, Milosevic M, McMillan A, Leschziner GD, Kumari V, Goadsby P, Simonds AK, Williams SC, Morrell MJ. Changes in Neurocognitive Architecture in Patients with Obstructive Sleep Apnea Treated with Continuous Positive Airway Pressure. EBioMedicine. 2016 May;7:221-9. doi: 10.1016/j.ebiom.2016.03.020. Epub 2016 Mar 25. PMID 27322475
- [Background] Xu H, Wang H, Guan J, Yi H, Qian Y, Zou J, Xia Y, Fu Y, Li X, Jiao X, Huang H, Dong P, Yu Z, Yang J, Xiang M, Li J, Chen Y, Wang P, Sun Y, Li Y, Zheng X, Jia W, Yin S. Effects of continuous positive airway pressure on neurocognitive architecture and function in patients with obstructive sleep apnoea: study protocol for a multicentre randomised controlled trial. BMJ Open. 2017 May 25;7(5):e014932. doi: 10.1136/bmjopen-2016-014932. PMID 28550021
- [Derived] Xu H, Liu Y, Li C, Li X, Shen L, Wang H, Liu F, Zou J, Xia Y, Huang W, Liu Y, Gao Z, Fu Y, Wang F, Huang S, Song Z, Song F, Gao Y, Peng Y, Zou J, Zhu H, Liu S, Li L, Zhu X, Xiong Y, Hu Y, Yang J, Li Y, Gao F, Guo Q, Huang H, Zhang W, Li J, Chen Y, Dong P, Yang J, Lv J, Wang P, Sun Y, Qian B, Yaffe K, Guan J, Yi H, Leng Y, Yin S. Effects of Continuous Positive Airway Pressure on Neuroimaging Biomarkers and Cognition in Adult Obstructive Sleep Apnea: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2025 Apr;211(4):628-636. doi: 10.1164/rccm.202406-1170OC. PMID 39998447